CLINICAL TRIAL: NCT07210281
Title: The Use of Ossein-hydroxyapatite Complex as an Adjunctive Treatment in Orthopedics and Traumatology
Brief Title: Osteogenon in Orthopedics and Traumatology
Acronym: Osteogenon
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Opole (Other)
Responsible Party: Principal Investigator, Piotr Morasiewicz, Professor, University of Opole
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-2025-003; P-2025-004 (Other Grant/Funding Number: University of Opole)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Patients With Fractures
Keywords: fractures; Osteogenon; ossein-hydroxyapatite complex; distal radius fractures; lower leg fracture; proximal humerus fractures
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteogenon (Experimental): received an ossein-hydroxyapatite complex
  Interventions: Drug: received an ossein-hydroxyapatite complex
- Control (No Intervention): did not receive an ossein-hydroxyapatite complex

INTERVENTIONS:
Drug: received an ossein-hydroxyapatite complex — Patients in the study group with fractures received an ossein-hydroxyapatite complex (830 mg of ossein-and-hydroxyapatite complex, with 444 mg of hydroxyapatite, equivalent to 178 mg of calcium and 82 mg of phosphorus) throughout the entire period following fracture healing. The tablets were taken orally, one tablet twice daily.
  Arms: Osteogenon

SUMMARY:
The aim of this study was to evaluate the supportive effect of the ossein-hydroxyapatite complex in fracture healing. The investigators hypothesized that the ossein-hydroxyapatite complex would positively impact fracture healing outcomes.The assessment covers clinical, radiological and biomechanical parameters.

DETAILED DESCRIPTION:
The role of ossein-hydroxyapatite complex in fracture healing requires further research.

The aim of the study was to evaluate the effect of ossein-hydroxyapatite complex (Osteogenon) as an adjunctive treatment on the outcome of conservative and surgical fractures treatment via comprehensive clinical, radiological and biomechanical assessments. The investigators aimed to reject the null hypothesis of the absence of beneficial effect of ossein-hydroxyapatite complex on fractures treatment outcomes. This would fill the existing gap in the scientific literature and enable a more widespread use of Osteogenon in the treatment of fractures in many trauma centers.

Patients in the study group with fractures received an ossein-hydroxyapatite complex (830 milligram [mg] of ossein-and-hydroxyapatite complex, with 444 mg of hydroxyapatite, equivalent to 178 mg of calcium and 82 mg of phosphorus) throughout the entire period following fracture healing. The tablets were taken orally, one tablet twice daily.

The drug Osteogenon used in our study had been approved for fracture treatment. The study was conducted in accordance with the Declaration of Helsinki and all applicable laws and regulations. All patients had provided their written informed consent and were informed of a voluntary nature of their participation in this study.

Patients participating in the study, both in the study and control groups, had to meet the inclusion criteria. The randomization method used was to evenly recruit the study and control groups as patients who met the inclusion criteria were recruited. Randomization took into account the equal distribution of gender and age in both groups.

Patients from both the experimental and control groups received the same recommendations regarding rehabilitation and had the same clinical and radiological follow-up protocol.

The following clinical, biomechanical and radiological parameters were assessed in the study: the period of immobilization, rate of bone union, analgesic use at the beginning of treatment, analgesic use during the follow-up, time to achieving pain relief, pain in 100 millimeter [mm] Visual Analogue Scale (VAS), number of patients declaring pain relief, rate of complications, time to resuming normal physical activity, grip strength, muscle strength during joint movement.

The period of immobilization was defined as the total number of days during which cast immobilization was maintained. The time to resuming normal physical activity was expressed in days and defined as the period from injury to return to work or school and normal everyday activities.

The rate of bone union was determined based on the percentage of patients who achieved clinical and radiological criteria of bone union. The radiological criteria of bone union were the presence of a minimum of 3 out of 4 consolidated cortical bone layers or trabecular transition between bone fragments on X-rays in 2 views. Clinical bone union was defined as the lack of pathological mobility, pain, or deformity during attempts to perform movements in the wrist area at the fracture site. Nonunion was defined as failure to meet the above criteria for 6 months after the fracture .

The investigators also assessed the number of patients on any analgesics (paracetamol, ibuprofen, non-steroidal anti-inflammatory drugs, tramadol) at the beginning of treatment and at the final follow-up. During regular follow-up visits, patients were asked about their pain intensity using the NRS (Numerical Rating Scale). A period of discontinuation of any pain medication was equivalent to a patient rating their pain level as 0 on the NRS. Time to achieving pain relief was expressed in days and defined as the period from the beginning to end of taking any analgesic drugs.

Complications were assessed based on medical and radiological records. The evaluated complications included nonunion, delayed bone union, fragment displacement, persistent pain, persistent swelling, limited range of motion, vascular damage, nerve damage, the need for revision surgery or repeated reduction and immobilization.

ELIGIBILITY:
Inclusion Criteria:

* no contraindications to taking Osteogenon
* a follow-up period of more than 3 months after treatment completion
* complete medical and radiological records
* a written informed consent
* not taking any other medications that could affect bone tissue remodeling
* not taking other medications that interact with Osteogenon
* no other limb pathologies (inflammatory or neurogenic)
* absence of comorbidities that could affect bone union

Exclusion Criteria:

* age under 18 years or over 85 years
* hypersensitivity to the active ingredient or to any of the excipients
* severe renal failure and dialysis therapy
* hypercalcemia
* hypercalciuria
* calcium-based kidney stones or tissue calcifications
* a follow-up period shorter than 3 months after treatment completion
* a lack of informed consent
* a lack of cooperation with the patient
* absent or incomplete medical and radiological records
* taking medications that could affect bone tissue remodeling
* taking medications that may interact with Osteogenon (e.g. thiazide diuretics)
* metabolic disorders
* post-traumatic skeletal deformities
* neuromuscular disorders
* post-inflammatory deformities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
period of bone union | at 6 months after randomisation
  assessed by data linkage to medical and radiological records
Achieving bone union | at 6 months after randomisation
  assessed by data linkage to medical and radiological records

SECONDARY OUTCOMES:
pain assessment | at 6 months after randomisation
  100mm Visual Analogue Scale (VAS)
  * 0 mm indicates "no pain"
  * 100 mm indicates "worst imaginable pain"
  * Higher scores on the VAS indicate a worse outcome (greater pain intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Marek Gierlotka, PROF, Study Chair — University of Opole
Locations (1):
- University Clinical Hospital in Opole, Opole, Opole Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
The data collected during our study are our own efforts and will be used to prepare our publications. Other authors are encouraged to conduct their own research.

REFERENCES:
- [Background] Morasiewicz P, Zaborska M, Sobczak M, Tomczyk L, Leyko P, Bobinski A, Kochanska-Bieri J, Pili D, Kazubski K. The Use of Osteogenon as an Adjunctive Treatment in Lower Leg Fractures. Pharmaceuticals (Basel). 2024 Nov 14;17(11):1531. doi: 10.3390/ph17111531. PMID 39598441
- [Background] Morasiewicz P, Zaborska M, Sobczak M, Tomczyk L, Pili D, Kazubski K, Leyko P. The Use of Ossein-Hydroxyapatite Complex in Conjunction with the Ilizarov Method in the Treatment of Tibial Nonunion. J Clin Med. 2025 May 12;14(10):3353. doi: 10.3390/jcm14103353. PMID 40429349